CLINICAL TRIAL: NCT03080233
Title: Validation of Clinical Decision Support Tool Information Technology Application for Stroke Diagnosis
Brief Title: Validation of Clinical Decision Support Tool for Acute Stroke Diagnosis (InstaDx)
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor, Aga Khan University
Other Study IDs: 4554-CHS-ERC-16
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Stroke, Acute
Keywords: stroke; Validation; Clinical decision support tool
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pakistani adult: Men and women aged 18 years or above,presenting with neurological deficit consistent with stroke in the Emergency Department at Aga Khan University Hospital
  Consenting to participate in the study

SUMMARY:
This is a observational validation study. The Stroke Clinical Decision Support Tool ( InstaDx) , an information technology application will be adapted and developed in accordance to evidence based clinical practice guidelines ( Level IA). Neurology Residents will be using the InstaDx CDST to improve their diagnostic accuracy and the findings will be validated against the review of a stroke subject expert. The study hypothesis is that Clinical Decision Support Tool used by neurology residents will have an agreement of >0.77 when compared to Stroke Expert (gold standard) in diagnosing type of ischemic stroke.

DETAILED DESCRIPTION:
Overall Objective: To adapt, develop and validate the clinical decision support tool, an information technology application to assist acute stroke diagnosis for use among neurology graduate trainees compared to stroke expert (gold standard).

Specific Aims:

1. To validate the adapted clinical decision support tool, an information technology application to assist acute ischemic stroke diagnosis for use among neurology residents compared to stroke expert (Gold standard) in the adult population presenting at a tertiary care hospital in Pakistan.

The study will be conducted in Emergency department and the Neurology ward at Aga Khan University Hospital. The data collector will enroll the patients meeting the eligibility criteria and providing informed consent. Neurology residents will use the Clinical Decision Support Tool application to assist in acute stroke diagnosis. In the second part, the Stroke Expert will independently assess all diagnosis. The purpose of this would be to validate the Clinical Decision Support Tool application to assist in acute stroke diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, >18 years of age.
2. Patients admitted with neurological deficit consistent with stroke.
3. Confirmation of stroke by objective modality of CT scan and MRI.
4. Consenting to participate in the study.

Exclusion Criteria:

1. Patients presenting with any type of Haemorrhagic stroke such as Sub-Arachnoid Haemorrhage, Intracerebral Haemorrhage and others.
2. Stroke due to any iatrogenic causes such as post-surgeries, trauma, or any rare or non atherosclerotic causes eg carotid dissection.
3. Patients signing LAMA (left against Medical Advice) and leaving undiagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men and women greater than or equal to 18 years of age presenting in emergency department with neurological deficit consistent with stroke, fulfilling our eligibility criteria and willing to give voluntary informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Validation_Primary Outcome Measure_ Sensitivity | Day 1
  Sensitivity of InstaDx used by Neurology Residents vs. Diagnosis by Stroke Expert
Validation_ Primary Outcome Measure_Specificity | Day 1
  Specificity of InstaDx used by Neurology Residents vs. Diagnosis by Stroke Expert
Validation_Primary Outcome Measure_Positive and Negative Predictive Values | Day 1
  Predictive Value of InstaDx used by Neurology Residents vs. Diagnosis by Stroke Expert

SECONDARY OUTCOMES:
Acceptability | Day 1
  Qualitative assessments by focus group discussion will be performed to incorporate user feedback

OTHER OUTCOMES:
Implementation Characteristics | Day 1
  Qualitative assessments by focus group discussion will be performed to evaluate the user feedback to further improve the uptake of the tool.

CONTACTS AND LOCATIONS:
Overall Officials: Ayeesha K Kamal, Principal Investigator — AKUH; Saadia S Choudhry, Principal Investigator — AKUH
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
This may be shared on request only.